CLINICAL TRIAL: NCT05909462
Title: Comparison of the Effects of Ultrasonography-guided Suprascapular Nerve Block and Intra-articular Shoulder Injection on Pain, Functional Status and Range of Motion in Patients With Adhesive Capsulitis; Randomized, Controlled Trial
Brief Title: Comparison of the Effects Suprascapular Nerve Block and Intra-articular Shoulder Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ayse Gulsen Dogan, Specialist Doctor, Hitit University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-56; Deniz İpek (Other: Hitit University); Mehmet Yalvaç (Other: Hitit University); Murat Doğan (Other: Hitit University); Abdulrahim Dündar (Other: Hitit University)
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; suprascapular nerve block; intra-articular shoulder injection; ultrasonography.
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Intervention Model Description: randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: double blind randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprascapular verve block (Experimental): 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine
  Interventions: Drug: 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine
- intraarticular shoulder injection (Experimental): 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine
  Interventions: Drug: 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine

INTERVENTIONS:
Drug: 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine — ultrasonography-guided suprascapular nerve block and intra-articular shoulder injection
  Other Names: intra-articular shoulder injection

SUMMARY:
Objectives: In this study, we aimed to compare the efficacy of ultrasonography-guided suprascapular nerve block and intra-articular shoulder injection treatment in terms of joint range of motion, pain and functional status in patients with adhesive capsulitis (AC).

Patients and Methods: 60 patients AC were included in our study. The patients were randomized into two groups according to the sealed envelope method. In the evaluation of the patients before the injection, age, gender, body mass index (BMI), occupation, education, duration of complaint, symptomatic side and dominant hand information were recorded. In the first group, 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine injection were mixed with the posterior approach method into the shoulder joint under the guidance of ultrasonography (USG). The second group underwent suprascapular nerve block (SSNB) injection with 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine under USG guidance. Shoulder range of motion (ROM), visual analog scale (VAS) scores and Shoulder Pain and Disability Index (SPADI) scores were compared before the injection, on the tenth day after the injection and at the third month after the injection.

Conclusion: As a result of our study, although it was observed that both methods provided improvement in the treatment process, the significant improvement in the SSNB group indicates that it is a more reliable treatment method in AC treatment.

DETAILED DESCRIPTION:
Sixty patients AC who applied to our Orthopedics-Traumatology and Physical Medicine-Rehabilitation Outpatient Clinic were included in our study. The study was approved by the Hitit University Clinical Research Ethics Committee (Decision number:2023-56). A well-informed written consent was obtained from all participants according to the principles of the Declaration of Helsinki. Patients with an age range of 18-65 years, adapting to the treatment program to be applied, diagnosed with unilateral stage 2-3 AC, no shoulder trauma in the last 3 months, no shoulder injections, no bleeding disorder, no history of malignancy, inflammatory disease and stroke were included in the study. The patients were randomized into two groups according to the sealed envelope method. In the evaluation of the patients before the injection, age, gender, body mass index (BMI), occupation, education, duration of complaint, symptomatic side and dominant hand information were recorded. Injections were made to the patients by the physiatrist and anesthetist researcher under the guidance of Logiq V2 portable USG device. In the first group, 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine injection were mixed with the posterior approach method into the shoulder joint under the guidance of USG. The second group underwent suprascapular nerve block injection with 2 ml of 40 mg triamcinolone acetonide and 4 ml of 1% lidocaine under USG guidance. In addition, pendulum and ladder-finger exercises were given to both groups as a home exercise program. Shoulder range of motion (ROM), visual analog scale (VAS) scores and Shoulder Pain and Disability Index (SPADI) scores were compared before the injection, on the tenth day after the injection and at the third month after the injection.

ELIGIBILITY:
Inclusion Criteria:

unilateral stage 2-3 AC

* no shoulder trauma in the last 3 months
* no shoulder injections
* no bleeding disorder
* no history of malignancy
* no history of inflammatory disease

Exlusion Criteria:

* malignancy
* inflammatory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in pain on The Shoulder Pain and Disability Index (SPADI) at the tenth day after the injection | baseline and on the tenth day after the injection
  SPADI is a valid and reliable questionnaire used in shoulder disorders. Possible scores range from 0 (no pain) to 100 (severe shoulder pain)= Changes tenth day after the injection-baseline
The effectiveness of suprascapular nerve block on pain is higher than intra-articular | between before treatment and on the tenth day after the injection
  Shoulder Pain and Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Comparison of the effects of ultrasonography-guided suprascapular nerve block and intra-articular shoulder injection on pain, functional status and range of motion in patients with adhesive capsulitis; randomized, controlled trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 21/01/2023-24/05/2023